CLINICAL TRIAL: NCT02147327
Title: Effects of Cord Blood 25-hydroxy-vitamin D Level on Early Neonatal Morbidities
Status: Completed | Type: Observational
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, birgul say, Fellow in Neonatology, Pediatrician, Zekai Tahir Burak Women's Health Research and Education Hospital
Other Study IDs: sevit25D3
Record Dates: First submitted 2014-05-21; First posted 2014-05-26 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Neonatal Hypocalcemia; Neonatal Sepsis
Keywords: vitamin D; cord blood; neonatal sepsis; neonatal morbidity
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cholecalciferol (vitamin D3) is a prohormone and its active form is 1,25 dihydroxycholecalciferol. This hormone has effect on both calcium, phosphorus and bone metabolism and also bone morrow, muscle, heart and immune system. For a long time, maternal low vitamin D level is a well known problem for our country and the level was reported as <10 ng/ml for 46-80% of mothers.The most prominent risk factor was determined as low socioeconomic status. Therefore, the level of 25-hydroxy-vitamin D is supposed to be in relation with several neonatal morbidities and maternal complications of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Term or preterm newborns which are hospitalized in the Neonatal Intensive Care Unit of our hospital

Exclusion Criteria:

* Preterm babies born before the 24. gestational week
* Babies with complex cardiac anomalies and/or dysmorphic features

Max Age: 30 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns which are hospitalized in the Neonatal Intensive Care Unit of our hospital
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
sepsis | 3 months but patients will be followed until discharge
feeding intolerance | 3 months but patients will be followed until discharge
hypocalcemia | 3 months but patients will be followed until discharge
bronchopulmonary dysplasia | 3 months but patients will be followed until discharge
patent ductus arteriosis | 3 months but patients will be followed until discharge
retinopathy of prematurity | 3 months but patients will be followed until discharge
maternal complications of pregnancy | from the beginning of gestation until birth process

SECONDARY OUTCOMES:
rachitism | 4 months but patients will be followed until discharge